CLINICAL TRIAL: NCT00773825
Title: Assessment of the Risk of Imprinting Defects in Children Born Following Assisted Reproductive Technologies (ART)
Brief Title: Genomic Imprinting and Assisted Reproductive Technologies
Acronym: EPIGEN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P040440
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Natural Pregnancy; Pregnancy, Ovarian
Keywords: Genomic imprinting; Reproductive techniques, assisted; Beckwith-Wiedemann syndrome; Angelman syndrome
MeSH Terms: conditions — Pregnancy, Ovarian; Helping Behavior; Beckwith-Wiedemann Syndrome; Angelman Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (serum, ADN) and placenta samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Pregnancy after ICSI or IVF
- 2: Pregnancy after ovarian stimulation
- 3: natural pregnancy

SUMMARY:
Genomic imprinting, referring to an epigenetic marking resulting in monoallelic gene expression, plays a critical role in development. Recently, various imprinting diseases were reported in animals (Large Offspring syndrome (LOS)) and humans (Beckwith-Wiedemann syndrome (BWS) and Angelman syndrome (AS)) born after ART. In all cases, an imprinting defect was involved (loss of methylation at ICR2 in BWS, at SNRPN in AS and at IGF2R DMR2 in LOS). These data suggest that ART procedures may impair the establishment or the maintenance (following fertilization) of methylation marks at maternally imprinted loci. In view of these data, the aim of this study is to determine if children born following ART exhibit an increased risk of imprinting defects. If the answer is yes, the second objective is to identify the problematic step in the ART procedure and thus to suppress or modify this step.

DETAILED DESCRIPTION:
Methodology: assessment of the methylation status at 9 different imprinted loci (using Southern blot and methyl-specific quantitative PCR) in 3 groups of patients: 150 children naturally conceived, 150 children conceived after ovarian stimulation but with in vivo fertilization, and 150 children conceived after ovarian stimulation and in VITRO fertilization. These analyses will be performed on cord blood. Fragments of placental tissue will also be collected for further analyses. Patients will be selected in maternity hospitals associated with ART departments ( ANTOINE BECLERE HOSPITAL, Cochin HOSPITAL, Saint-Vincent de Paul HOSPITAL, Jean VERDIER HOSPITAL, Tenon HOSPITAL and Dijon Hospital).

This work is also a unique opportunity to establish a DNA, RNA and tissue collection allowing further investigation regarding other epigenetic modifications than DNA methylation, not only at imprinted loci, but also in other genomic regions regulated by epigenetic modifications.

ELIGIBILITY:
Inclusion Criteria:

Mother :

* Age: 26 to 40 at conception
* Single foetus pregnancy
* Signed informed consent
* Affiliation to French health benefits
* Absence of maternal pathology
* Normal foetal karyotype (if available)
* Known procedure of ovarian stimulation
* ART procedure without sperm or oocyte donation
* ART in a participating ART departments
* Delivery in a participating hospital

Father

* Age : 18 to 50 at conception
* Signed informed consent

Exclusion Criteria:

* Abnormal foetal karyotype (if available)
* Delivery before 35 weeks of amenorrhea
* Delivery in not participating hospital
* Delivery complication leading to the absence of sample collection

Ages: 26 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women followed in a participating ART departments
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2007-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the methylation status at 9 imprinted loci in cord blood collected just after birth. | At the birth

SECONDARY OUTCOMES:
Assessment of other epigenetic marks (histone modifications) at imprinted loci and at non imprinted but epigenetically regulated loci. | At the birth

CONTACTS AND LOCATIONS:
Overall Officials: Yves Le BOUC, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Trousseau Hospital, Paris, France

REFERENCES:
- [Background] Gicquel C, El-Osta A, Le Bouc Y. Epigenetic regulation and fetal programming. Best Pract Res Clin Endocrinol Metab. 2008 Feb;22(1):1-16. doi: 10.1016/j.beem.2007.07.009. PMID 18279777
- [Background] Rossignol S, Steunou V, Chalas C, Kerjean A, Rigolet M, Viegas-Pequignot E, Jouannet P, Le Bouc Y, Gicquel C. The epigenetic imprinting defect of patients with Beckwith-Wiedemann syndrome born after assisted reproductive technology is not restricted to the 11p15 region. J Med Genet. 2006 Dec;43(12):902-7. doi: 10.1136/jmg.2006.042135. Epub 2006 Jul 6. PMID 16825435
- [Background] Gicquel C, Gaston V, Mandelbaum J, Siffroi JP, Flahault A, Le Bouc Y. In vitro fertilization may increase the risk of Beckwith-Wiedemann syndrome related to the abnormal imprinting of the KCN1OT gene. Am J Hum Genet. 2003 May;72(5):1338-41. doi: 10.1086/374824. No abstract available. PMID 12772698
- [Background] Gaston V, Le Bouc Y, Soupre V, Burglen L, Donadieu J, Oro H, Audry G, Vazquez MP, Gicquel C. Analysis of the methylation status of the KCNQ1OT and H19 genes in leukocyte DNA for the diagnosis and prognosis of Beckwith-Wiedemann syndrome. Eur J Hum Genet. 2001 Jun;9(6):409-18. doi: 10.1038/sj.ejhg.5200649. PMID 11436121